CLINICAL TRIAL: NCT04563130
Title: Use of Cryocompression to Reduce Chemotherapy-induced Peripheral Neuropathy in Gynecologic Cancer: a Randomized Controlled Trial
Brief Title: Cryocompression to Reduce Chemotherapy-induced Peripheral Neuropathy in Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00106236
Record Dates: First submitted 2020-09-16; First posted 2020-09-24 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Gynecologic Cancer; Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryocompression (Experimental): Patients will be randomized to receive cryocompression on one hand and foot using ice bags and compression socks.
  Interventions: Behavioral: Cryocompression
- Control (No Intervention): Patients will be randomized to receive no intervention on the opposite hand and foot.

INTERVENTIONS:
Behavioral: Cryocompression — Cryocompression will be administered using ice bags and compression socks/ surgical gloves
  Arms: Cryocompression

SUMMARY:
The aim of this study is to evaluate the effect of cryocompression therapy on the incidence and degree of taxane-induced peripheral neuropathy in gynecologic cancer patients receiving chemotherapy. Subjects will serve as their own controls, and will be randomized to cryocompression therapy on their dominant versus non-dominant hand and foot, with standard of care treatment (no intervention) on the opposite hand and foot. Compression therapy will be performed using commercially available compression socks and disposable surgical gloves, and cryotherapy will be achieved by applying bags of ice to the compression devices. Subjects will complete baseline neuropathy surveys including the Patient Neurotoxicity Questionnaire (PNQ) and the Functional Assessment of Cancer Therapy (FACT) -Taxane (FACT-NTX), which includes the sensory subscale of the FACT-NTX. Subjective symptoms will be assessed at baseline, before each cycle of chemotherapy and cryocompression, and one month after completion of 6 cycles. In addition, tactile sensation will be assessed with the monofilament test at baseline and one month after completion of 6 cycles of chemotherapy and cryocompression. The primary outcomes are the proportion of patients with PNQ grade C or higher and decline in tactile sensitivity from baseline based on the monofilament test. The investigators hypothesize that cryocompression will reduce chemotherapy-induced peripheral neuropathy in patients with gynecologic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Gynecologic cancer diagnosis (ovarian, cervical, endometrial cancer; adenocarcinomas of likely primary gynecologic origin based on cytology or FNA in conjunction with radiologic impression will be eligible)
* Plan to receive at least 6 cycles of paclitaxel administered every 3 weeks at Duke Cancer Institute. Patients receiving neoadjuvant chemotherapy with a plan for interval debulking will be eligible.
* ECOG performance status of 0-1
* Latex allergy does not exclude a subject from the study. Non-latex gloves will be provided.

Exclusion Criteria:

* Treated with prior neurotoxic chemotherapeutic agents
* Baseline diagnosis of peripheral neuropathy such as diabetic neuropathy, or associated with conditions including but not limited to fibromyalgia, cryoglobulinemia and Raynaud's disease.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Change in Patient Neurotoxicity Questionnaire [PNQ] (patient reported assessment) over time | baseline, after each dose of paclitaxel and cryocompression, and one month after completion of chemotherapy.
  PNQ is a patient-reported questionnaire that consists of 2 items, representing motor and sensory components, with increasing grades for worsening symptoms. Patients will respond to each question for each of their 4 extremities by grading sensory and motor symptoms as A (no neuropathy), B (mild neuropathy), C (moderate neuropathy that does not interfere with activities of daily living [ADL]), D (moderate neuropathy that does interfere with ADL), or E (severe neuropathy that interferes with ADL). The first primary outcome of this study is the proportion of patients with Patient Neurotoxicity Questionnaire (PNQ) grade C or higher peripheral sensory neuropathy any time after the baseline assessment.
Change in Semmes-Weinstein monofilament test (tactile disturbance) over time | baseline, one month after completion of chemotherapy.
  The monofilament test is a simple, inexpensive test to assess tactile sensation and detect peripheral sensory neuropathy. Tactile perception is assessed at 10 locations on the hand and 10 locations on the foot. Patients who exhibit any decline in tactile sensitivity in response to light touch from baseline to completion of taxane treatment will be counted as events for the primary outcome assessment.

SECONDARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy (FACT) -Taxane [FACT-NTX] (patient reported assessment) over time | baseline, after each dose of paclitaxel and cryocompression, and one month after completion of chemotherapy.
  The FACT-NTX is a patient self-reported 11-item questionnaire used for evaluating symptoms and concerns specifically associated with chemotherapy induced neuropathy. The total score ranges from 0-44, and a lower FACT-NTX score corresponds to worsening neuropathy. For both the FACT-NTX and the sensory subscale of the FACT-NTX, a significant decrease in the score is defined as a decrease exceeding 10% from baseline.
Tolerability of cryocompression: scale | after each dose of paclitaxel and cryocompression
  Subjects will be asked to complete a cryocompression tolerability assessment after each chemotherapy session in which they will answer the question, "How tolerable was the cryocompression procedure for you?" on a scale from 0 to 100. A score of 0 means "not tolerable at all" and a score of 100 is "very tolerable". Pain, abnormal sensation, and adherence to cryocompression will also be evaluated as patient-reported measures of tolerability.
Acceptability: scale | immediately after the intervention
  Subjects will be asked to complete a cryocompression acceptability assessment after each chemotherapy session in which they answer the questions, "How acceptable was the cryocompression procedure to you?" and "How likely are you to continue with cryocompression at your next chemotherapy treatment?" on a scale from 0 to 100, with 0 being "not acceptable, not likely to continue" and 100 being "very acceptable, very likely to continue".

CONTACTS AND LOCATIONS:
Overall Officials: Laura Havrilesky, MD, MHSc, Principal Investigator — Duke University Hospital
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anastasio MK, Unnithan S, Scott A, Hayes T, Shah S, Moss HA, Erkanli A, Havrilesky LJ. Cryocompression to Reduce Peripheral Neuropathy in Gynecologic Cancer: A Randomized Controlled Trial. Obstet Gynecol. 2023 Dec 1;142(6):1459-1467. doi: 10.1097/AOG.0000000000005419. Epub 2023 Oct 26. PMID 37883997